CLINICAL TRIAL: NCT03728946
Title: Interscalene Block With and Without Liposomal Bupivacaine in Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orthopaedic & Neurosurgery Specialists (Other)
Responsible Party: Principal Investigator, Paul Sethi, Principal Investigator, Orthopaedic & Neurosurgery Specialists
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018016
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Rotator Cuff Tear; Postoperative Pain
MeSH Terms: conditions — Rotator Cuff Injuries; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liposomal Bupivacaine Interscalene Block (Experimental): Liposomal bupivacaine anesthetic will be administered as an interscalene block during rotator cuff repair surgery and total shoulder arthroplasty.
  Interventions: Drug: Liposomal Bupivacaine
- Bupivacaine Interscalene Block (No Intervention): Bupivacaine anesthetic will be administered as an interscalene block during rotator cuff repair surgery and total shoulder arthroplasty.

INTERVENTIONS:
Drug: Liposomal Bupivacaine — Addition of 15mL of liposomal bupivacaine to 15mL of standard nerve block anesthetic solution containing 0.5% bupivacaine and 4mg of decadron
  Other Names: EXPAREL
  Arms: Liposomal Bupivacaine Interscalene Block

SUMMARY:
The purpose of this study is to examine the difference in perioperative pain after shoulder surgery with a standard bupivacaine nerve block compared to liposomal bupivacaine enhanced nerve block alone in TSA and ARCR. Data will be compared using VAS scores and opiate consumption between the two groups. The hypothesis of this study is that an interscalene nerve block with liposomal bupivacaine will decrease both postoperative VAS pain scores and total narcotic consumption when compared to a standard bupivacaine interscalene nerve block alone.

DETAILED DESCRIPTION:
Arthroscopic rotator cuff repair (ARCR) and shoulder arthroplasty (TSA) provide excellent clinical outcomes but are often associated with significant postoperative pain, frequently managed with oral opioid medication. Orthopedic surgeons prescribe approximately 32 unused pills per shoulder surgery and are the third largest prescribers of opiates in the USA. It is incumbent upon the orthopedic community to identify postoperative pain management methods which reduce the need for narcotic medication following shoulder procedures as a means to mitigate the impact of orthopedic procedures on this epidemic.

The use of intraoperative local and regional anesthesia or field blocks, in conjunction with multimodal pharmacological strategies, is an accepted approach for managing surgical pain and reducing opiate use but requires peer reviewed protocols to gain wider acceptance.

Interscalene nerve block with bupivacaine remains a gold standard for peri-operative analgesia, but is associated with significant rebound pain due to the short duration of the local anesthetics. Recent studies have demonstrated that the addition of a liposomal bupivacaine field block may lower pain and enhance patient satisfaction throughout the first postoperative week. Liposomal bupivacaine has recently received FDA approval for ISB, but the data regarding its efficacy in nerve blocks is sparse.

The purpose of this pilot study is to determine if liposomal bupivacaine-enhanced interscalene nerve blocks can be used to improve peri-operative pain control methods, limit narcotic use, and provide appropriate postoperative analgesia compared to standard bupivacaine blocks. Primary and secondary outcome measures will be collected as number of opiates taken and self-reported VAS pain scores over a 14 day postoperative period, respectively.

The hypothesis of this study is that an interscalene nerve block with liposomal bupivacaine will decrease both postoperative VAS pain scores and total narcotic consumption when compared to a standard bupivacaine interscalene nerve block alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 undergoing rotator cuff repair or total shoulder arthroplasty

Exclusion Criteria:

* Pregnant
* Documented drug of alcohol abuse
* Active narcotic use prior to surgery
* Neurological deficit
* Allergy to amide anesthetics
* Not cleared by primary care physician
* Hydrocodone or oxycodone intolerance
* Enrollment in another clinical trial or past cognitive or mental health status that interferes with study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Opiate Consumption | Post-operative days 1-14
  Total amount of narcotics consumed during the postoperative period, measured in morphine equivalents (OME)

SECONDARY OUTCOMES:
VAS Pain Scores | Post operative days 1-14
  A standardized measure of subjective pain on a scale of 0 to 10, from zero pain to excruciating pain, respectively
Likert Pain Satisfaction Rating | Post operative days 1-14
  A standardized measure of patient satisfaction with pain management from 1 (very unsatisfied) to 5 (very satisfied)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Greenwich Hospital, Greenwich, Connecticut
  - Orthopaedic & Neurosurgery Specialists, Greenwich, Connecticut
  - Stamford Ambulatory Surgical Center, Stamford, Connecticut
  - Atlantis Orthopaedics, Atlantis, Florida
  - Atlantis Orthopaedics, Palm Beach Gardens, Florida
  - Southern Oregon Orthopedics, Inc., Medford, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar K, Gulotta LV, Dines JS, Allen AA, Cheng J, Fields KG, YaDeau JT, Wu CL. Unused Opioid Pills After Outpatient Shoulder Surgeries Given Current Perioperative Prescribing Habits. Am J Sports Med. 2017 Mar;45(3):636-641. doi: 10.1177/0363546517693665. Epub 2017 Feb 9. PMID 28182507
- [Background] Lee CY, Robinson DA, Johnson CA Jr, Zhang Y, Wong J, Joshi DJ, Wu TT, Knight PA. A Randomized Controlled Trial of Liposomal Bupivacaine Parasternal Intercostal Block for Sternotomy. Ann Thorac Surg. 2019 Jan;107(1):128-134. doi: 10.1016/j.athoracsur.2018.06.081. Epub 2018 Aug 28. PMID 30170012
- [Background] Pedoto A, Amar D. Liposomal Bupivacaine for Intercostal Nerve Block: Pricey or Priceless? Semin Thorac Cardiovasc Surg. 2017 Winter;29(4):538-539. doi: 10.1053/j.semtcvs.2017.08.016. Epub 2017 Aug 30. No abstract available. PMID 28967536
- [Background] Rice DC, Cata JP, Mena GE, Rodriguez-Restrepo A, Correa AM, Mehran RJ. Posterior Intercostal Nerve Block With Liposomal Bupivacaine: An Alternative to Thoracic Epidural Analgesia. Ann Thorac Surg. 2015 Jun;99(6):1953-60. doi: 10.1016/j.athoracsur.2015.02.074. Epub 2015 Apr 23. PMID 25912739
- [Background] Surdam JW, Licini DJ, Baynes NT, Arce BR. The use of exparel (liposomal bupivacaine) to manage postoperative pain in unilateral total knee arthroplasty patients. J Arthroplasty. 2015 Feb;30(2):325-9. doi: 10.1016/j.arth.2014.09.004. Epub 2014 Sep 16. PMID 25282071
- [Background] Vandepitte C, Kuroda M, Witvrouw R, Anne L, Bellemans J, Corten K, Vanelderen P, Mesotten D, Leunen I, Heylen M, Van Boxstael S, Golebiewski M, Van de Velde M, Knezevic NN, Hadzic A. Addition of Liposome Bupivacaine to Bupivacaine HCl Versus Bupivacaine HCl Alone for Interscalene Brachial Plexus Block in Patients Having Major Shoulder Surgery. Reg Anesth Pain Med. 2017 May/Jun;42(3):334-341. doi: 10.1097/AAP.0000000000000560. PMID 28157791